CLINICAL TRIAL: NCT07255859
Title: CRYSTALSIGHT: Clinical Evaluation of OCCUTRACK's CRYSTALSIGHT Device Through Remote Monitoring for Disease Recurrence of Wet Aged-Related Macular Degeneration Using Eye Gaze Tracking (Cohort 2.0).
Brief Title: CRYSTALSIGHT Cohort 2.0
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Laude Augustinus, Senior Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-3705
Record Dates: First submitted 2025-06-23; First posted 2025-12-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Maculopathy
Keywords: aged-related macular degeneration; diabetic macular edema; diabetic retinopathy; choroidal neovascularization; wet aged-related macular degeneration; gaze tracking; dry aged-related macular degeneration; maculopathy
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Choroidal Neovascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amsler Grid (Active Comparator): The Amsler grid is a tool used to monitor the macula, the central part of the retina, for changes in vision that can be indicative of various eye conditions, particularly age-related macular degeneration (AMD). It helps detect and monitor metamorphopsia (distorted vision) or scotoma (blind spots) in the central visual field.
  Interventions: Diagnostic Test: Amsler Grid
- CRYSTALSIGHT Arm (Experimental): OCCUTRACK's CRYSTALSIGHT device tracks these eye movements with generated patterns on the screen, a visual assessment of affected and unaffected eyes is achieved without expensive optics and at home on any tablet or laptop computer.
  CRYSTALSIGHT is a home-based gaze-tracking readily available for home hyperacuity monitoring for these and other high-risk eyes with diagnosed wet-AMD.
  Interventions: Device: CRYSTALSIGHT

INTERVENTIONS:
Diagnostic Test: Amsler Grid — The Amsler grid is a tool used to monitor the macula, the central part of the retina, for changes in vision that can be indicative of various eye conditions, particularly age-related macular degeneration (AMD). It helps detect and monitor metamorphopsia (distorted vision) or scotoma (blind spots) in the central visual field.
  Arms: Amsler Grid
Device: CRYSTALSIGHT — OCCUTRACK's CRYSTALSIGHT device tracks these eye movements with generated patterns on the screen, a visual assessment of affected and unaffected eyes is achieved without expensive optics and at home on any tablet or laptop computer.
  CRYSTALSIGHT is a home-based gaze-tracking readily available for home hyperacuity monitoring for these and other high-risk eyes with diagnosed wet-AMD.
  Arms: CRYSTALSIGHT Arm

SUMMARY:
Age-Macular Degeneration (AMD) is a common eye condition and a leading cause of vision loss among people age 50 and older. It causes damage to the macula, a small area near the centre of the retina needed for sharp, central vision. It is estimated that the prevalence of early and late AMD in Asian populations aged 40 to 79 were 6.8% and 0.56% respectively. Prevalence in white populations estimated from large population studies were 8.8% and 0.59% respectively. With the aging population and people living longer, these numbers will only increase. Hence, this study aims to develop a system to evaluate OCCUTRACK's CRYSTALSIGHT device through remote monitoring for disease recurrence of wet aged-related macular degeneration using eye gaze tracking.

DETAILED DESCRIPTION:
Age-Related Macular Degeneration (AMD) and Diabetic macular Edema (DME) is one of the main causes of central vision loss. Most patients require pharmacologic treatment with anti-vascular endothelial growth factor (VEGF) agents with multiple follow-up visits that include optical coherence tomography (OCT), visual acuity testing and multiple injections.

The high frequency of visits puts pressure on eye clinics and can be extremely stressful for both patients and their caregivers. Therefore, portable and rapidly deployable self-administered home-based examination devices are key to making telemedicine a reality.

OCCUTRACK Medical Solutions has developed a portable, self-administered device designed for gaze-tracking and monitoring of patients with retinal diseases such as AMD and DME, and choroidal neovascularization (CNV) that require multiple anti-VEGF injections.

The team have confirmed the performance of the CRYSTALSIGHT device and validated the retinal thickness measurements obtained with this device by comparing it to in-hospital Optical Coherence Tomography (OCT) (Heidelberg Spectralis). In this study, the team will conduct a randomized clinical trial RCT to compare the efficacy and cost-effectiveness of a Pro Re Nana (PRN) management regimen enhanced with the CRYSTALSIGHT home monitoring device for the detection of central metamorphopsia with existing PRN standard of care for patients with AMD or DME exiting the anti-VEGF injection regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects in the age group ≥ 55 to 99 years old.
2. Both genders
3. Able to understand verbal spoken instructions in British/American English, Chinese or Bahasa Melayu and demonstrate device functionality and implementation.
4. Able to turn on and connect the CRYSTALSIGHT device to a computer independently or with the help of family.
5. Subjects undergoing treatment for Wet-AMD without any signs and symptoms of recurrence of active AMD (AMD recurrence: choroidal neovascularisation, intraretinal or subretinal fluid is present) with OCT lesion fluid volume more than 2 mm2 or ILM height more than 300µm.
6. Ability to comply with the study protocol, in the investigator's judgment.
7. Subjects must be able to understand and provide informed consent. A signed informed consent form must be provided before any study assessments.

Exclusion Criteria:

1. Unable to understand verbal spoken instructions and demonstrate device functionality and implementation.
2. Unable to turn on and connect the CRYSTALSIGHT device to a computer independently.
3. Any ocular surgery in the previous 3 months, or vitrectomy in the previous 12 months
4. Any history of macular pathology unrelated to AMD affecting vision or contributing to the presence of intraretinal or subretinal fluid in the study eye
5. Any concurrent intraocular condition in the study eye that, in the opinion of the investigator, could either reduce the potential for visual improvement or require medical or surgical intervention during the study
6. Any prior or concomitant treatment for CNV or vitreomacular-interface abnormalities in the study eye.
7. History of idiopathic or autoimmune-associated uveitis in either eye
8. Active ocular inflammation or suspected or active ocular or periocular infection in either eye.

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy Using One-Sided Confidence Interval or One-Sided Hypothesis Test | 12 Months
  To assess whether the CRYSTALSIGHT device is non-inferior to the standard of care (Amsler grid) in detecting recurrence of wet-AMD during patient recall, by comparing both generated scores, validated by OCT readings.

SECONDARY OUTCOMES:
Correlation with Optical Coherence Tomography (OCT) | 12 Months
  To determine the correlation between CRYSTALSIGHT gaze scores and average OCT height readings
User Experience & Functionality | 12 Months
  Qualitative assessment of usability and patient adherence to the home testing protocol will be conducted by evaluating completion rates of CRYSTALSIGHT testing twice weekly. Consistent compliance will be interpreted as an indicator of protocol feasibility and user-friendliness, suggesting that the testing procedure was sufficiently accessible and manageable for patients to maintain regular adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Augustinus Laude, MBChB, MSc, FRCSEd (Ophth), FA, Principal Investigator — Tan Tock Seng Hospital; Zheng Kuang Noel Soh, BSc, Study Director — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT07255859/Prot_000.pdf